CLINICAL TRIAL: NCT00440713
Title: Phase 3 Study of Aripriprazole in the Treatment of Post-Traumatic Stress Disorder Symptoms
Brief Title: Aripiprazole in the Treatment of Post-Traumatic Stress Disorder Symptoms
Acronym: AripipPTSD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2007-02-22; First posted 2007-02-27 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Depression; Anxiety; Efficacy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aripiprazole
Behavioral: Interpersonal Therapy

SUMMARY:
32 outpatients with a Posttraumatic Stress Disorder were included in a randomized comparative single-blind study to study the efficacy of aripiprazole to treat post-traumatic stress symptoms.

The hypothesis is that aripiprazole has an efficacy to reduce PTSD symptoms

DETAILED DESCRIPTION:
All patients which agreed to participate and signed the informed consent, were interviewed to be enrolled if they filled the inclusion and exclusion criteria.

The inclusion criteria were: both genders, aged 18 to 60, diagnosis of PTSD DSM-IV criteria by a trained psychiatrist after the application of the SCID-I. Women must be using contraceptive methods during the study. Women had to be using contraceptive methods during the study. The exclusion criteria were to have a diagnostic of the following conditions: schizophrenic disorder, delusional disorder, bipolar disorder, psychotic depression episode and psychoactive substance dependency disorder in the previous 6-month period, instable medical diseases, and pregnancy.

All included patient was submitted at baseline to a socio-demographic inventory and to a psychometric evaluation, the latter were reapplied at weeks 8 and 16. The psychometric evaluation consist of self-report instruments: CAPS to measure PTSD symptoms severity, the Beck Depression Inventory (BDI) [29] and the Beck Anxiety Inventory (BAI) [30] to measure the depressive and the anxiety symptoms severity, the Medical Outcome Scale short form (MOS-SF-36) [31] and the Social adjustment scale (SAS) [32] to evaluate quality of life and social adjustment. A 7.5mg single dose of aripiprazole was prescribed, and the patient was evaluated each two weeks and dose could be increased or decreased depending of their tolerability to side effects. After 16-week the drug was discontinued over a two week period.

Thirty-two outpatients were included after filling the inclusion and exclusion criteria. Twenty-four (75%) were women and 8 (25%) men. Eighteen (56.3%) were married, eight (25%) single, and six (18.7%) were widowed or divorced. Their mean age was 38.41 (+/-10.97) years old, and the mean time since trauma happened was 50.87 (+/-77.21) months. Three (9.4%) patients have been victims of sexual abuse, four (12.5%) kidnapped, four (12.5%) held hostage in prison rebellion, 7 (21.88%) lost a close person to homicide, 8 (18.75%), suffered a homicide attempt.

Nine (28%) patients discontinued the treatment before the second assessment. Six (18.7%) patients discontinued the medication because of adverse events (anxiety, psychomotor agitation, nausea, and insomnia), three (3) patients abandoned the treatment and we lost contact with them. Six (6) patients had at least a second assessment, but did not complete 16-week trial, three due to a complete remission and a resistance to continue on the study and three discontinued due to lack of clinical improvement. The BDI baseline mean score from the dropouters was 28.7 (+/- 12.7) higher compared to the completers 25 (+/- 11.2) showing a statistically significant difference (t=.2167 p<.02) The mean dose was 9.6 (+/-4.3) mg/day, with the dose range of 3.75 to 15 mg day.

An intention-to-treat analysis using the Last Observation Carried Forward (LOCF) including the baseline outcome data found a CAPS mean score at baseline of 82.7 (+/- 23.1) and 51.4 (+/-31.4) on endpoint, over 38% reduction from the baseline. Comparing the data using the t test the difference between before and after the treatment was statistically significant (t=.000002, p<.001 - Table and Graph 1).

When using a concept of 30% decrease at CAPS mean score from baseline as a response to treatment, 17 (53.1%) patients have a response, and when using a more restrictive concept of 50% decrease at CAPS mean score 13 (40.6%) patients responded to the treatment.

The mean BAI score at baseline was 31.7 (+/- 13.4) and at the end-point were 25.4 (+/-18.2) (t=.01, p<.05) The SAS mean index score at baseline was 2.4 (+/-.45) and on the endpoint 2.27 (+/- .57) (t=.033, p<.05). The SF-36 mean score at baseline was 76.6 (+/-14.11) and at baseline 94.01 (+/- 25.06) (t=.0006, p<.05). On all measures, excepted on BDI, the differences between baseline and endpoint means were statistically significant. On the BDI with a mean score at baseline of 26.06 (+/- 11.6) and at the end-point of 21.35 (+/-12.6), the difference wasn't statistically significant (t=.58, p<.05).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PTSD (after SCID-I application by a trained psychiatrist).
* Use of an effective contraceptive method when the subject is women with sexual activity and with risk of pregnancy.

Exclusion Criteria:

* Clinical diagnosis of schizophrenic, delusional, psychotic depression, schizoaffective, bipolar or borderline personality (after SCID-I application by the a trained psychiatrist).
* Clinical diagnosis of psychoactive substance dependence within 6-months before the study enrollment.
* To have decompensated medical diagnostics needing urgent treatment
* being pregnant.
* using psychoactive drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2004-01; Study Completion 2006-03

PRIMARY OUTCOMES:
CAPS (Clinician Administered Posttraumatic Scale) score (PTSD symptoms)

SECONDARY OUTCOMES:
Beck Depression Inventory
Beck Anxiety Inventory
Social Adjustment Scale
Global Assessment Functioning
MOS SF-36, quality of life
Dropout
complete the trial

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo F Mello, M.D., Principal Investigator — Federal University of São Paulo